CLINICAL TRIAL: NCT01089387
Title: Intracavernous Bone Marrow Stem-cell Injection for Post Prostatectomy Erectile Dysfunction
Acronym: INSTIN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT06-07; 2008-A01248-47 (Other: Afssaps)
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2011-04

CONDITIONS: Prostate Cancer; Erectile Dysfunction
Keywords: radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- injection of bone marrow cells (Experimental)
  Interventions: Biological: injection of bone marrow mononucleated cells

INTERVENTIONS:
Biological: injection of bone marrow mononucleated cells — Four different concentration of BMMNC will be tested in four groups of 3 patients. In group 5 (n=19): one cell concentration corresponding to the best dose determined by analysis of the previous groups will be tested.
  Other Names: cell therapy

SUMMARY:
Erectile dysfunction is a frequent adverse event after radical prostatectomy for prostate cancer.

It is the consequence of penile vascular damage, mainly arterial insufficiency and venous leakage associated with fibrosis of the corpus cavernous. Apoptosis of penile cells, including mesenchymal cells, smooth muscle cells and endothelial is believed to play an important role in the pathophysiology of post prostatectomy erectile dysfunction.

Bone marrow mononucleated cells (BMMNC) contain different cell types that may replace the damaged penile cells after radical prostatectomy. These are mainly: mesenchymal stem cells, endothelial progenitor cells and hematopoietic stem cell. Intracavernous injection of BMMNC may therefore find application in the treatment of post prostatectomy erectile dysfunction.

The aims of this phase I-II study is to test the safety of autologous intracavernous BMMNC injection and to evaluate benefit for the patient concerning recovery of natural erection. Patients with penile vascular abnormality (echo-doppler) and localized prostate cancer (considered as cured by radical prostatectomy) will be included in this study.

Four different doses of BMMNC will be tested.

DETAILED DESCRIPTION:
We have shown in a rat model of post prostatectomy erectile dysfunction that BMMNC injection replace apoptotic cavernous cells and restore erectile function.

In the pig, the injection of high dose of BMMNC into the corpus cavernosus does not cause side effect. Moreover, the BMMNC remains at the injection site.

ELIGIBILITY:
Inclusion Criteria:

* Localized prostate cancer: PSA (Prostate Specific Antigen) prior to radical prostatectomy < 10 ng/ml, histopathologic analysis of the prostate showing a prostate cancer with Gleason score ≤ 7, negative margin, absence of effraction of the prostatic capsule, pT1 or pT2 N0 or NX.
* PSA=0 ng/ml 6 months after radical prostatectomy.
* Normal erectile function prior to radical prostatectomy.
* Penile arterial insufficiency and or venous leakage (doppler) at the time of inclusion: PSV <25 cm/sec, PSV >25 cm/sec, EDV>5cm/sec, RI<0,75.

Exclusion Criteria:

* Non localized prostate cancer.

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Absence of serious adverse event (general or local) | 6 months
  Side effects envisaged: priapism, local inflammation after cell injection

SECONDARY OUTCOMES:
Recovery of natural erection, improvement of penile doppler parameters | 6 month
  Evaluation of erectile recovery using validated quesitonnaires (IIEF15, EHS, UCLA-PCI)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Henri Mondor-Albert Chenevier-Centre Intercommunal de Créteil, Créteil, France

REFERENCES:
- [Result] Yiou R, Hamidou L, Birebent B, Bitari D, Le Corvoisier P, Contremoulins I, Rodriguez AM, Augustin D, Roudot-Thoraval F, de la Taille A, Rouard H. Intracavernous Injections of Bone Marrow Mononucleated Cells for Postradical Prostatectomy Erectile Dysfunction: Final Results of the INSTIN Clinical Trial. Eur Urol Focus. 2017 Dec;3(6):643-645. doi: 10.1016/j.euf.2017.06.009. Epub 2017 Jun 24. PMID 28753830
- [Result] Yiou R, Hamidou L, Birebent B, Bitari D, Lecorvoisier P, Contremoulins I, Khodari M, Rodriguez AM, Augustin D, Roudot-Thoraval F, de la Taille A, Rouard H. Safety of Intracavernous Bone Marrow-Mononuclear Cells for Postradical Prostatectomy Erectile Dysfunction: An Open Dose-Escalation Pilot Study. Eur Urol. 2016 Jun;69(6):988-91. doi: 10.1016/j.eururo.2015.09.026. Epub 2015 Oct 4. PMID 26439886
- [Derived] Khera M, Albersen M, Mulhall JP. Mesenchymal stem cell therapy for the treatment of erectile dysfunction. J Sex Med. 2015 May;12(5):1105-6. doi: 10.1111/jsm.12871. No abstract available. PMID 25974235